CLINICAL TRIAL: NCT03930914
Title: Vagus Nerve Stimulation in Treatment of Postural Orthostatic Tachycardia Syndrome
Acronym: POTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Dysautonomia International (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 10415
Record Dates: First submitted 2019-04-08; First posted 2019-04-29 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Postural Orthostatic Tachycardia Syndrome
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Treatment to Sham (Other): Subjects randomized to the sequence Active Treatment/Sham Treatment arm will be instructed to first use the Parasym (TM) TENS device as active treatment for the first phase of the study. Next, they will be instructed to use the Parasym (TM) TENS device as sham treatment for the second phase of the study.
  Interventions: Device: Parasym (TM) Transcutaneous Electrical Nerve Stimulation (TENS) Device
- Sham to Active Treatment (Other): Subjects randomized to the sequence Sham Treatment/Active Treatment arm will be instructed to use the Parasym (TM) TENS device as sham treatment for the first phase of the study. Next, they will be instructed to use the Parasym (TM) TENS device as active treatment for the second phase of the study.
  Interventions: Device: Parasym (TM) Transcutaneous Electrical Nerve Stimulation (TENS) Device

INTERVENTIONS:
Device: Parasym (TM) Transcutaneous Electrical Nerve Stimulation (TENS) Device — Daily use of Parasym (TM) device on tragus or ear lobe, as assigned treatment arm

SUMMARY:
Postural orthostatic tachycardia (POTS) is characterized by abnormalities in the autonomic nervous system in the body. The autonomic nervous system controls and regulates body functions such as heart rate, breathing, digestion, and more.

The investigator has shown that patients with POTS have higher cardiovascular and adrenergic activating autoantibodies (AAb), which likely changes the normal make-up of POTS. There are autoantibodies that have been suggested by a few reports of their presence in POTS, but their role different aspects of POTS is unknown. The study will look at the body's responses in patients with POTS. The crossover study design is to have half of the patients will start with sham followed by active stimulation and half will start by active followed by sham stimulation. It is anticipated that results will provide a potential therapeutic approach based on the understanding of POTS.

ELIGIBILITY:
Inclusion Criteria:

-Female or male participants age 18-80

Group 1 (20 participants):

* A physician-based diagnosis of POTS
* Participants that have a postural pulse rise of >35 for adolescents and >30 for adults with a Blood Pressure (BP) that does not drop >10/5 mmHg will be qualified. These participants may be on salt and fluid loading.

Group 2 (10 participants):

* Previously diagnosed with POTS
* Patients is on Intravenous immunoglobulin (IVIG) infusion but who have an incomplete symptomatic response

Exclusion Criteria:

* Age < 18 years
* Sick sinus syndrome, 2nd or 3rd degree Atrioventricular (AV) block, bifascicular block or prolonged 1st degree AV block (PR>300ms).
* Currently pregnant women or women planning on becoming pregnant ≤ 6 months
* History of hypotension due to autonomic dysfunction
* Have a secondary causes of tachycardia (acute anemia or blood loss, drugs, significant cardiomyopathy, diabetes mellitus)
* Patients with active implants (such as a cardiac pacemaker, or a cochlear implant).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2021-12-07 (Actual)

PRIMARY OUTCOMES:
Average change in orthostatic heart rate | 2 and 4 months
  We will measure the average change in heart rate between supine and standing using continuous ECG after two and four months of daily vagal nerve stimulation
Long term effects on M2 muscarinic autoantibody levels | 2 and 4 months
  The average change in M2 muscarinic autoantibody levels measured from blood specimens obtained after two and four months of daily vagal nerve stimulation.
Long term effects on beta 1-adrenergic autoantibody levels | 2 and 4 months
  The average change in beta 1-adrenergic autoantibody levels measured from blood specimens obtained after two and four months of daily vagal nerve stimulation.
Long term effects on alpha 1-adrenergic autoantibody levels | 2 and 4 months
  The average change in alpha 1-adrenergic autoantibody levels measured from blood specimens obtained after two and four months of daily vagal nerve stimulation.
Average change in heart rate variability | 2 and 4 months
  We will measure the average change in heart rate variability based on 5 minute ECG after two and four months of daily vagal nerve stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Xichun Yu, MD, Principal Investigator — University of Oklahoma; Stavros Stavrakis, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No